CLINICAL TRIAL: NCT00173849
Title: The Role of SDF-1/CXCR4 in Metastasis of Oral Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700656
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Oral Cancer
Keywords: oral cancer; CXCR4; stromal-cell-derived factor-1(SDF-1); metastasis
MeSH Terms: conditions — Mouth Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
Investigate the role of SDF-1/CXCR4 in the metastasis of oral squamous cell carcinoma

DETAILED DESCRIPTION:
Oral cancer is the most common head and neck malignancy, constituting near 9% of all cancers (1). Squamous cell carcinoma (SCC) is the most common histopathologic type of the oral malignancies, accounting for more than 90% of cancers occurring in this region (2). The presence or absence of regional lymph node metastases is the single most important factor affecting prognosis in patients with oral cancer. Cure rates for oral cancer are decreased by approximately 50 percent in patients having cervical lymph node metastasis (3).

Tumor metastasis is the hallmark of malignancy, and is probably a result of the interaction between tumor cells and a supportive microenvironment. Malignant cells that have the capability to metastasize to a particular organ may have various properties supporting their tissue invasion or growth such as enhanced adherence to the microvascular cells of the organ, higher responsiveness to chemotactic signals released from the target organs and increased response to local soluble or tissue associated growth signals in the target organ (4,5). Though there are several molecules expressed or produced in cancer cells are considered the metastatic factors, it remains unknown which factors produced by the lymph node or tissue affect the metastasis of cancer cells.

Chemokines are a large family of pro-inflammatory polypeptide cytokines, consisting of small (7-15 kDa), structurally related heparin-binding proteins. They are grouped into CXC chemokines and CC chemokines, on the basis of the characteristic presence of four conserved cysteine residues (6-8). Chemokines are produced locally in the tissues and act on target cells through G-protein-coupled receptors, which are characterized structurally by seven transmembrane spanning domains. Chemokines are involved in the attraction and activation of mononuclear and polymorphonuclear leukocytes to sites of inflammatory responses, bacterial or viral infections, allergy, cardiovascular diseases and wound healing (4, 8-13). Chemokines are known to also function as regulatory molecules in the leukocyte maturation, trafficking, and homing of T and B lymphocytes, in the development of lymphoid tissues, and in dendritic cell maturation (14,15). Other functions of chemokines have been described more recently, particularly for the CXC chemokines. The role of chemokines in malignant tumors is not clear yet. Some chemokines may enhance innate or specific host immunity against tumor dissemination. On the other hand, some may advocate tumor growth and metastasis by promoting tumor cell proliferation, migration or angiogenesis in tumor tissue (4). Reports have suggested that several types of cancer, such as breast (16), ovary (17), prostate (18), kidney (19), brain (20), lung (21), and thyroid (22), expressed the chemokine receptor and used the chemokines to metastasize to the target organ as in the homing of hematopoietic cells.

SDF-1 belongs to the CXC chemokine family and is a ligand for CXCR4 (23, 24). SDF-1 was initially cloned by Tashiro et al. (25) and later identified as a growth factor for B cell progenitors, a chemotactic factor for T cells and monocytes, and in B-cell lymphopoiesis and bone marrow myelopoiesis (23, 26-27). Most of the chemokine receptors interact with pleural ligands, and vice versa, but the SDF-1/CXCR4 receptor ligand system has been shown to involve a one-on-one interaction (28, 29). Recently, several studies have been conducted to detect the mRNA expression of CXCR4 and SDF-1 in solid tumors. The results are not uniform, and the relevance to cancer progression is not determined (30, 31). Sehgal et al. (30, 32) concluded that CXCR4 plays an important role of proliferation and tumorigenic properties of human glioblastoma tumors. Muller et al. (33) have reported that SDF-1 signaling through CXCR4 interaction appears to determine the directional migration of breast cancer cells through the basement membrane. Furthermore in vivo, the interaction between SDF-1 and CXCR4 significantly represses the metastatic potential of breast cancer cells to lymph node and lung. Barnard and his colleagues (34, 35) showed the contrary results that CXCR4 mRNA expression was reduced in hepatocellular carcinoma tissue when compared with noncancerous tissue, but was not changed in colon, esophageal, and gastric cancer. They also found reduced mRNA expression of SDF-1 in these malignant tissues (31). Thus, there is a diversity of views on the role of the SDF-1/CXCR4 receptor ligand system in malignant tissues. And such studies are limited in oral cancer.

Since metastasis of oral cancer occur frequently through the lymphatic system, and metastasis is a key prognostic factor for the disease. Evaluation of the relationship between SDF-1/CXCR4 system and metastasis in oral cancer could help us understand whether this system is important in the metastasis of this disease.

We hypothesized that SDF-1/CXCR4 (ligand/receptor) system plays an important role in oral cancer metastasis. To test this hypothesis, we will investigate (1) the distribution of CXCR4 protein expression in cancer and lymph node tissues by means of immunohistochemical analysis of tissue samples obtained from surgical operation, (2) the relationship between CXCR4 expression and clinicopathological findings with special reference to cancer metastasis, (3) the expression of SDF-1 and CXCR4 in the cancer cell lines cells and tissues, (4) the chemotactic activity and the growth-promoting effect of SDF-1 on cancer cell lines cells, (5) the role of Src, MAPK, and Akt signal transduction pathway in this response, (6) the effect of the blocking agent on this response.

Undoubtedly, the findings of this study will help us understand whether SDF-1/CXCR4 system could be a focal point of anti-cancer research. If oral SCC that express high levels of CXCR4 show a consistently higher incidence of lymphatic and distant metastasis, then blocking SDF-1/CXCR4 signaling may be a novel approach to inhibit metastasis in these patients. The development of SDF-1/CXCR4 system antagonists will provide opportunity to improve the survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Oral squamous cell carcinoma

Exclusion Criteria:

* other pathological type

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ting Tan, MD, PhD, Principal Investigator — National Taiwan University Hospita;
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan